CLINICAL TRIAL: NCT01826253
Title: Observational Study of Oxygen Delivery During a Fractional Fluid Expansion
Acronym: OR
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Principal Investigator, Marc-Olivier FISCHER, Medecine Doctor, University Hospital, Caen
Other Study IDs: A12-D37-VOL.13
Record Dates: First submitted 2013-03-20; First posted 2013-04-08 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2013-05

CONDITIONS: Hypovolemia; Impaired Oxygen Delivery; Cardiac Output, Low
Keywords: Hypovolemia; Fluid challenge; Fluid expansion; Oxygene delivery; Cardiac output
MeSH Terms: conditions — Hypovolemia; Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hypovolemia: Fluid expansion
  Interventions: Drug: hydroxyethylstarch 130/0.4

INTERVENTIONS:
Drug: hydroxyethylstarch 130/0.4 — Bolus of 100ml of HES 130/0.4 repeated until maximization of cardiac output

SUMMARY:
Fluid expansion during cardiocirculatory insufficiency was helped by cardiac output monitoring. However, the goal of fluid expansion was to increase the oxygen delivery, which consider cardiac output, but also Haemoglobin which decrease during a fluid challenge. The maximalization of cardiac output could decrease the oxygen delivery if the haemodilution was too wide. The aim of this study was to describe the oxygen delivery during a fluid expansion conducted for cardiac output maximalization, following actual guidelines.

DETAILED DESCRIPTION:
One group of 20 anticipated patients

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years
* Patients in intensive care after cardiac surgery under mechanically ventilation and with oesophageal Doppler

Exclusion Criteria:

* Arrythmia
* Pregnancy or childrens
* Patients without cardiac output monitoring with oesophageal Doppler
* Patients without medical indication for fluid expansion
* Urgency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated patients after elective cardiac surgery with oesophageal Doppler for cardiac output monitoring and arterial and venous central line
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Measurement of oxygen delivery | only during the fluid challenge
  Retrospective calculation of oxygen delivery (ml.min.m-2)during a fractional fluid expansion every 100ml of hydroxyethyl starch until cardiac output maximalization with oesophageal Doppler and arterial gazes (for PaO2 and Haemoglobin)from arterial line.

SECONDARY OUTCOMES:
Study of central venous saturation | only during the fluid challenge
  Central venous gazes after each mini fluid challenge until cardiac output maximalization, from a central line

OTHER OUTCOMES:
study of cerebral and muscular oxygenation measured with near-infrared spectroscopy | only during the fluid challenge
  study of cerebral and muscular oxygenation measured with near-infrared spectroscopy after each mini fluid challenge until cardiac output maximalization, from a central line

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Caen, Caen, France